CLINICAL TRIAL: NCT03481517
Title: The Interest of Wound Infiltration With Local Anesthetic Agent for Laparoscopic Appendectomy in Adult: a Double Blind, Prospective, Randomized Control Trial
Brief Title: Wound Infiltration With Local Anesthetic Agent for Laparoscopic Appendectomy in Adult
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201710064RINB
Record Dates: First submitted 2018-02-01; First posted 2018-03-29 (Actual); Last update posted 2020-04-27 (Actual); Status verified 2020-04

CONDITIONS: Appendicitis Acute
Keywords: adult; appendectomy; appendicitis; local anesthesia; pain
MeSH Terms: conditions — Appendicitis; Pain | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wound with local anesthesia (Experimental): 5 mL Bupivacaine is injected into subcutaneous area near surgical wound
  Interventions: Drug: Bupivacaine
- Wound without local anesthesia (No Intervention): Nothing is injected into subcutaneous area near surgical wound

INTERVENTIONS:
Drug: Bupivacaine — Bupivacaine 5 mL subcutaneous injection to surgical wound during operation.
  Other Names: Marcaine
  Arms: Wound with local anesthesia

SUMMARY:
Acute appendicitis is one of the most common acute abdomens that need surgical intervention. Laparoscopic surgery much decreases postoperative pain of wound, however, pain remains an important determinant of recovery after surgery. Intraoperative local anesthetic agent infiltrated locally into surgical wound to relieve postoperative pain is a feasible and safe method suggested in some literature. However, there is no routine use of this method in clinical practice because its benefit is still unknown. Besides, very few evidence could be found in literature review. To date, there is still no double blinded, prospective, randomized control trial addressing in evaluation of its interest. In this study, the investigators aim at investigating the benefit of wound infiltration with local anesthetic agent (bupivacaine) for laparoscopic appendectomy in adult. The study design is a double blind, prospective, randomized control trial with a 1:1 allocation ratio. Fifty adult patients with appendicitis will be included. The control group undergo laparoscopic appendectomy without wound infiltration with local anesthetic agent, the intervention group undergo laparoscopic appendectomy with wound infiltration with local anesthetic agent intraoperatively. The clinical characteristics, outcomes, and patient's satisfaction will be recorded and analyzed. The investigators hope this study can provide a high level evidence in pain management of patient undergo laparoscopic surgery.

ELIGIBILITY:
Including criteria:

1. Clinical diagnosis of appendicitis and undergo laparoscopic appendectomy
2. Age more than 20 years
3. Well comprehensive in speaking Chinese

Exclusion criteria:

1. Age no more than 20 years
2. Pregnancy
3. Can not cooperate with evaluation
4. Convert to open surgical method, resect more organs than appendix
5. Using patient control analgesia
6. Allergy to local anesthetic agent

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2018-04-23 (Actual); Primary Completion 2019-07-08 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Pain score of surgical wound of the patient | within 24 hours after surgery
  Using Visual Analog Score (from 0 to 10, 0 indicate no pain and 10 indicate maximal pain) to evaluate pain of surgical wound of the patient

SECONDARY OUTCOMES:
Satisfaction of the patient | up to one month after surgery
  Using questionnaire to evaluate satisfaction of the patient about surgery and hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Yang Hsiao, M.D., Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan